CLINICAL TRIAL: NCT00002201
Title: Safety and Efficacy of Ritonavir (ABT-538) in Combination With Nelfinavir in HIV-Infected Subjects.
Brief Title: A Study of Ritonavir (ABT-538) When Used With Nelfinavir in HIV-Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 245D; M96-581
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; HIV Protease Inhibitors; Ritonavir; Nelfinavir; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir; Nelfinavir

INTERVENTIONS:
Drug: Ritonavir
Drug: Nelfinavir mesylate

SUMMARY:
The purpose of this study is to see if it is safe and effective to give ritonavir plus nelfinavir to HIV-infected patients. This study will also see how ritonavir and nelfinavir are absorbed by the body and how they affect the level of HIV in the blood.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Documentation of a positive ELISA test for HIV confirmed by immunoblot, or a positive HIV RNA test using the Roche PCR assay, or the Chiron bDNA assay.
* HIV RNA measurement of > 5,000 copies/ml within 3 weeks of baseline visit.
* Signed, informed consent from parent or legal guardian for patients less than 18 years of age.
* Access to a refrigerator for storing study drug.

Prior Medication:

Allowed:

Anti-HIV therapy other than protease inhibitor therapy.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Evidence of acute infection, as measured by vital signs, physical examination, 12-lead electrocardiogram and laboratory assessments.
* Condition that may obscure the proper observation of the safety or activity of the treatment regimens.

Concurrent Medication:

Excluded:

* Midazolam, alprazolam, clorazepate, diazepam, estazolam, flurazepam, triazolam, zolpidem, quinidine, amiodarone, encainide, flecainide, propafenone, bepridil, terfenadine, astemizole, cisapride, bupropion, clozapine, rifabutin, meperidine, propoxyphene, piroxicam, pimozide, ergotamine, dihydroergotamine, and rifampin.
* Anti-retroviral therapy initiated prior to study entry.
* Any other medication, including over-the-counter medicine and alcohol, taken without the permission of the primary investigator.

Patients with the following prior conditions are excluded:

* History of significant drug hypersensitivity.
* History of psychiatric illness that would preclude compliance with the protocol.
* Prior enrollment in this study.

Prior Medication:

Excluded:

* Investigational drugs within 30 days prior to drug administration.
* Prior treatment with licensed or investigational HIV protease inhibitor.

  1. Active substance abuse.
* Positive urine screen for recreational drugs. NOTE:
* The presence of cannabis is not exclusionary unless the investigator believes its use will interfere with patient compliance.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Hosp, Baltimore, Maryland, United States

REFERENCES:
- [Background] Raines CP, Flexner C, Sun E, Heath-Chiozzi M, Lewis RH, Fields C, Deetz C, Apuzzo L, Eshleman SH, Jackson JB, Gallant JE. Safety, tolerability, and antiretroviral effects of ritonavir-nelfinavir combination therapy administered for 48 weeks. J Acquir Immune Defic Syndr. 2000 Dec 1;25(4):322-8. doi: 10.1097/00042560-200012010-00005. PMID 11114832